CLINICAL TRIAL: NCT07031999
Title: Use of Biocompatible Thermoplastic Impregnated With Vancomycin as a Temporary Orthopedic Spacer
Acronym: ORTOPLA
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hospital Universitario Evangelico de Curitiba (Other)
Collaborators: Pontifícia Universidade Católica do Paraná (Other)
Responsible Party: Principal Investigator, Felipe Francisco Bondan Tuon, Professor, Hospital Universitario Evangelico de Curitiba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ORTOPLA; PUCPR (Other: PUCPR)
Record Dates: First submitted 2025-06-09; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Implant Failure; Infection
Keywords: PLA; prosthesis
MeSH Terms: conditions — Infections

STUDY DESIGN:
Intervention Model Description: The interventional group include the use of articular spacer with antibiotic.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PLA spacer (Experimental): PLA spacer implantation
  Interventions: Combination Product: PLA spacer

INTERVENTIONS:
Combination Product: PLA spacer — This is a phase 1/2 prospective, interventional, non-randomized, single-arm clinical study designed to evaluate the safety of using temporary articular spacers printed in PLA (polylactic acid) impregnated with vancomycin in patients with periprosthetic infections of the hip, knee, or shoulder.

SUMMARY:
With the progressive aging of the population and the rising number of individuals with degenerative diseases, there has been an increasing indication for joint replacement arthroplasties as a treatment for osteoarthritis in major joints. Knee, hip, and shoulder prostheses have become effective treatment options for joint degeneration, aiming to restore motor function, improve mobility, and relieve pain. In this context, infection remains a major concern, as it can lead to implant removal and the need to replace it with a temporary implant (articular spacer) combined with local antibiotic delivery and systemic antimicrobial therapy-both essential for the complete resolution of the infectious condition.

Polylactic acid (PLA) is a biocompatible and biodegradable polymer that can be used in 3D printing technologies to develop customized implants and temporary spacers for the treatment of periprosthetic and bone infections, in addition to its potential application in bone reconstruction. The development of such products through reverse engineering, combined with advanced imaging techniques and specialized computational systems, enables the creation of patient-specific implant models, thus optimizing the recovery process.

Therefore, this research project proposes the development and application of a polymer with suitable antimicrobial activity, based on reverse engineering and 3D printing technologies, for the design of orthopedic prostheses and implants. This study aims to address treatment needs in Brazil, where the cost of bone substitutes and articular spacers remains high, especially in orthopedic reconstruction, and where public healthcare systems face challenges in providing adequate and affordable solutions.

In this sense, the development of customized, biocompatible, low-cost, and antimicrobial implants may have a significant impact on both patient outcomes and the public health system. This technology is innovative, as it will bring a novel category of medical product to the national market with potential for global reach, thereby representing a substantial advancement in the healthcare field.

ELIGIBILITY:
Inclusion Criteria:

* Age:

Patients aged 18 years or older.

Gender:

Individuals of all genders are eligible for participation.

Indication for Prosthesis Replacement:

Patients with an active infection related to a hip, knee, or shoulder prosthesis who require implant removal due to infection and placement of an antibiotic-loaded spacer.

Informed Consent:

Patients or their legal guardians must have signed the Informed Consent Form (ICF), authorizing their participation in the study.

Active Infection:

Patients must present with clinical signs of active periprosthetic infection, such as pain, fever, or purulent discharge at the implant site.

Willingness for Follow-Up:

Patients must be willing to attend outpatient follow-up visits and undergo clinical evaluations over a 6-month postoperative period.

Exclusion Criteria:

* Inactive Infection:

Patients without signs of active prosthetic infection (i.e., no fistula, purulent discharge, or erythema).

Pregnancy or Lactation:

Pregnant or breastfeeding women.

Severely Compromised Immunosuppression:

Patients with conditions that significantly impair the immune system, including:

Solid organ or hematopoietic stem cell transplantation.

Untreated HIV infection or CD4 count < 350 cells/mm³.

Prolonged use of immunosuppressive therapy (e.g., corticosteroids at doses equivalent to >0.5 mg/kg/day of prednisone for more than 3 weeks).

Clinically Incompatible Conditions:

Patients with severe or unstable medical conditions that may compromise procedural safety or the ability to adhere to study follow-up.

Inability to Attend Postoperative Follow-Up:

Patients unable to comply with postoperative follow-up visits or telephone consultations due to mobility restrictions or lack of access.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Control of periprosthetic infection | From enrollment to the end of treatment at 6 months post-implantation
  Measured Variable:
  Rate of complications or adverse events, including implant misfit, residual infection, implant rejection, and other adverse outcomes such as wound dehiscence or seroma.
  Definition:
  Implant misfit will be defined as the inability of the spacer to properly adapt to the prosthetic defect site, as assessed intraoperatively by the orthopedic surgeon. Residual infection will be characterized by the persistence of clinical signs of infection following spacer implantation (e.g., fistulas, purulent discharge).
  Analysis Metric:
  Proportion of patients who experienced any adverse event (e.g., number of patients with residual infection, implant misfit, or other complications).
  Aggregation Method:
  Proportion of patients presenting at least one adverse event (e.g., proportion of patients with implant misfit or residual infection).
  Time Point for Analysis:
  Assessment following spacer implantation, with follow-up extending up to 6 months post-implantation.

SECONDARY OUTCOMES:
Surgical complications | From enrollment to the end of treatment at 6 months post-implantation
  Measured Variable:
  Rate of periprosthetic infection control, defined as the absence of infection signs following spacer implantation.
  Definition:
  Infection control will be considered achieved when no clinical signs of infection are present (e.g., fever, persistent pain, purulent discharge) by the final evaluation point.
  Analysis Metric:
  Proportion of patients with complete infection control within 6 months after spacer implantation.
  Aggregation Method:
  Proportion of patients with successful infection eradication.
  Time Point for Analysis:
  Monthly follow-up visits for 6 months post-surgery.
  Evaluator:
  Clinical evaluation will be performed by the orthopedic surgeon during outpatient visits, supported by laboratory tests (when necessary) to confirm infection eradication.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tuon FF, Cieslinski J, Ono AFM, Goto FL, Machinski JM, Mantovani LK, Kosop LR, Namba MS, Rocha JL. Microbiological profile and susceptibility pattern of surgical site infections related to orthopaedic trauma. Int Orthop. 2019 Jun;43(6):1309-1313. doi: 10.1007/s00264-018-4076-7. Epub 2018 Aug 2. PMID 30069593